CLINICAL TRIAL: NCT02034682
Title: The Effect of Hydroxyethylstarch 6% 130/0.4 in a Balanced Electrolyte Solution (Volulyte®) Compared to Gelatine (Geloplasma®) on Microvascular Reactivity and Tissue Oxygen Saturation During Haemodilution Measured With Near-infrared Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/1085; 2013-005209-30 (EudraCT Number)
Record Dates: First submitted 2013-12-11; First posted 2014-01-13 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Microvascular Reactivity; Tissue Oxygen Saturation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volulyte 6% (Experimental): - Volulyte 6% (HES 130/0.4 in an isotonic composition). In 1000 ml:
  * Maize starch 60 gr. Molar substitution 0.38-0.45. 130000 Da
  * Na acetate trihydrate 4.63 gr
  * Sodium Chloride 6.02 gr
  * Potassium Chloride 0.3 gr
  * MgCl 0.3 gr
  * Sodium hydroxide-hydrochloric acid & H2O
  Interventions: Drug: Volulyte 6%
- Geloplasma (Active Comparator): In 1000 ml:
  * Modified fluid gelatin 30 gr
  * Sodium Chloride 5.4 gr
  * Potassium Chloride 0.37 gr
  * MgCl 0.14 gr
  * Sodium lactate 3.36 gr
  Interventions: Drug: Geloplasma

INTERVENTIONS:
Drug: Volulyte 6% — During elective coronary artery bypass grafting surgery, patients need to be attached to a cardiopulmonary bypass circuit. Administration of Volulyte 6% to the cardiopulmonary bypass circuit.
  Arms: Volulyte 6%
Drug: Geloplasma — During elective coronary artery bypass grafting surgery, patients need to be attached to a cardiopulmonary bypass circuit. Administration of Geloplasma to the cardiopulmonary bypass circuit.
  Arms: Geloplasma

SUMMARY:
The aim of this study is to compare 6% hydroxyethyl starch (HES) 130/0.4 in a balanced electrolyte solution (Volulyte®) with modified fluid gelatin (Geloplasma®) as the priming solution for the cardiopulmonary bypass (CPB) circuit. The microvascular reactivity and the effects on tissue (StO2) and cerebral (ScO2) oxygen saturation will be examined using near-infrared spectroscopy (NIRS).

ELIGIBILITY:
Inclusion Criteria:

Adult consenting patients scheduled for elective coronary artery bypass grafting surgery on moderately hypothermic (> 32°C) CPB without blood transfusion. Age ≥ 18 years.

Exclusion Criteria:

Exclusion criteria are an ejection fraction < 25%, a known allergy to HES, admission of HES or gelatines within the preceding 2 weeks, renal insufficiency (creatinine > 2.0 mg/dl), significant hepatic disease (liver function tests > 3x upper limit of normal), history of cerebrovascular disease, significant carotid artery stenosis (> 60%), perioperative use of corticosteroids, and need for vasopressor or inotropic therapy before surgery. An expected haematocrit on CPB, calculated based on preoperative haematocrit, calculated blood volume and amount of cardioplegia, of < 23% is also considered an exclusion criterium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Value of the StO2 recovery slope (recStO2) after postocclusive ischaemia. | after 3 minutes of postocclusive ischaemia
  Values are measured, using near-infrared spectroscopy.

SECONDARY OUTCOMES:
Change of values of ScO2 during cardiopulmonary bypass (CPB ). | Continuously during cardiopulmonary bypass (= maximum 3 hours).
Change of value of StO2 during cardiopulmonary bypass. | Continuously during cardiopulmonary bypass(= maximum 3 hours).
Change of blood gas analyses during cardiopulmonary bypass. | Continuously during cardiopulmonary bypass(= maximum 3 hours).
Change of haemodynamics during cardiopulmonary bypass. | Continuously during cardiopulmonary bypass(= maximum 3 hours).
Urinary output during cardiopulmonary bypass. | At the end of cardiopulmonary bypass(= after maximum 3 hours)..
Use of vasoactive medication during cardiopulmonary bypass. | During complete cardiopulmonary bypass(= maximum 3 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Moerman, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

REFERENCES:
- [Derived] Vandenbulcke L, Lapage KG, Vanderstraeten KV, De Somer FM, De Hert SG, Moerman AT. Microvascular reactivity monitored with near-infrared spectroscopy is impaired after induction of anaesthesia in cardiac surgery patients: An observational study. Eur J Anaesthesiol. 2017 Oct;34(10):688-694. doi: 10.1097/EJA.0000000000000684. PMID 28834795
- See also: Related Info — http://www.uzgent.be